CLINICAL TRIAL: NCT00088452
Title: Childhood Absence Epilepsy Rx PK-PD-Pharmacogenetics Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: U01NS045911 (NIH); U01NS045803 (NIH)
Record Dates: First submitted 2004-07-26; First posted 2004-07-27 (Estimated); Results first posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2017-02

CONDITIONS: Childhood Absence Epilepsy; Petit Mal Epilepsy; Epilepsy; Seizures
Keywords: childhood absence epilepsy; CAE; petit mal epilepsy; epilepsy; seizures; ethosuximide; lamotrigine; valproic acid
MeSH Terms: conditions — Epilepsy, Absence; Epilepsy; Seizures | interventions — Ethosuximide; Lamotrigine; Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ethosuximide (Active Comparator): Ethosuximide
  Frequency and Duration: twice a day, every day for the duration of the study treatment
  Formulation: Two formulations were used (actual formulation used was dependent on the patient's weight and ability to swallow): 250mg Zarontin capsules OR 250 mg/5 mL Zarontin syrup
  Dosing: Ethosuximide was titrated in predetermined increments every 1-2 weeks during a 16-week titration period. The titration continued until the patient a) achieved seizure freedom by clinical and EEG criteria, b) reached the maximal allowed study drug dose, c) reached the maximal tolerated dose, or d) developed dose-exiting criteria (treatment failure), whichever came first. Maximum allowed dose: 60 mg/kg/day or 2000 mg/day (whichever was lower)
  Interventions: Drug: Ethosuximide
- Lamotrigine (Active Comparator): Lamotrigine
  Frequency and Duration: twice a day, every day for the duration of the study treatment
  Formulation: Three formulations were used (actual formulation used was dependent on the patient's weight): 5mg Lamictal chewable tablets OR 25 mg Lamictal chewable tablets OR 25 mg (Lamictal tablets
  Dosing: Lamotrigine was titrated in predetermined increments every 1-2 weeks during a 16-week titration period. The titration continued until the patient a) achieved seizure freedom by clinical and EEG criteria, b) reached the maximal allowed study drug dose, c) reached the maximal tolerated dose, or d) developed dose-exiting criteria (treatment failure), whichever came first. Maximum allowed dose: 12 mg/kg/day or 600 mg/day (whichever was lower).
  Interventions: Drug: Lamotrigine
- Valproic acid (Active Comparator): Valproic acid
  Frequency and Duration: twice a day, every day for the duration of the study treatment
  Formulation: Two formulations were used (actual formulation used was dependent on the patient's weight): 250mg Depakote capsules OR 125mg Depakote sprinkles.
  Dosing: Depakote was titrated in predetermined increments every 1-2 weeks during a 16-week titration period. The titration continued until the patient a) achieved seizure freedom by clinical and EEG criteria, b) reached the maximal allowed study drug dose, c) reached the maximal tolerated dose, or d) developed dose-exiting criteria (treatment failure), whichever came first. Maximum allowed dose: 60 mg/kg/day or 3000 mg/day (whichever was lower)
  Interventions: Drug: Valproic acid

INTERVENTIONS:
Drug: Ethosuximide — Ethosuximide is a common treatment for childhood absence epilepsy.
  Other Names: Zarontin
  Arms: Ethosuximide
Drug: Lamotrigine — Lamotrigine is a common treatment for childhood absence epilepsy.
  Other Names: Lamictal
  Arms: Lamotrigine
Drug: Valproic acid — Valproic acid is a common treatment for childhood absence epilepsy.
  Other Names: Depakote
  Arms: Valproic acid

SUMMARY:
The purpose of this study is to determine the best initial treatment for childhood absence epilepsy.

DETAILED DESCRIPTION:
Childhood absence epilepsy (CAE) is a common pediatric epilepsy syndrome that affects 10 to 15 percent of all children with epilepsy. Individuals with CAE have brief staring spell seizures that occur suddenly, unpredictably, and frequently throughout the day. These seizures impair the children's ability to learn and play, and lead to higher injury rates.

There are many medications used to treat seizures, but only 3 generally are used as the first treatment for children with CAE: ethosuximide, lamotrigine, and valproic acid. The goal of this study is to determine which of these 3 medicines is the best first choice as treatment for children with CAE.

Approximately 439 children, recruited over a 3-year period at 32 medical centers in the US, will take part in this 5-year study. Participants will be randomly given one of the 3 common CAE treatments-ethosuximide, lamotrigine, or valproic acid-and will make regular visits to a clinic every 1 to 3 months for approximately 2 years. During the visits, participants will undergo regular testing to determine if the medicine is working, to watch for side effects, and to help researchers learn more about the responses to these medicines. In addition, researchers hope to develop methods that may be used in the future to help choose the best medicine for each individual diagnosed with CAE.

Also included in the study will be pharmacokinetics and pharmacogenetics research. Pharmacokinetics is the study of how the body absorbs, distributes, metabolizes, and excretes drugs. Pharmacogenetics is the study of genetic determinants of the response to drugs. Knowledge gained from this study may lead to individualized treatment for children with CAE, and may also be beneficial for other pediatric and adult seizure disorders.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Clinical diagnosis of Childhood Absence Epilepsy consistent with the International League against Epilepsy Proposal for Revised Classification of Epilepsies and Epileptic Syndromes (3).
* EEG: Interictal EEG demonstrating bilateral synchronous symmetrical approximate 3 Hz spike waves on a normal background with at least one burst lasting >/= (greater than or equal to) 3 seconds.
* Age > 2.5 years and < 13 years of age at study entry.
* Body weight >/= (greater than or equal to) 10 kilograms.
* Body Mass Index: BMI for age =/< 99th percentile (based on the CDC BMI for age growth curves for boys/girls [http://www.cdc.gov/growthcharts], Appendix 1).
* Hepatic:
* AST/ALT < 2.5 times the upper limit of normal
* Total bilirubin < 1.5 times the upper limit of normal.
* Hematologic:
* Absolute neutrophil count >/= (greater than or equal to) 1500/mm3.
* Platelets >/= (greater than or equal to) 120, 000 /mm3.
* Female subjects must be premenarchal at the time of enrollment and must be willing to practice abstinence for the duration of the study.
* Parent/legal guardian(s) willing to sign an IRB approved informed consent.
* Subject assent (when appropriate and as dictated by local IRB).

Exclusion Criteria:

* Treatment for CAE with anti-seizure medications (AED) for a period of greater than 7 days prior to randomization.
* History of a major psychiatric disease (e.g., psychosis, major depression).
* History of autism or pervasive development disorder.
* History of non-febrile seizures other than typical absence seizures. This includes a history of an afebrile generalized tonic clonic seizure.
* Clinical signs and symptoms consistent with a diagnosis of juvenile absence epilepsy or juvenile myoclonic epilepsy as delineated by the International League against Epilepsy Proposal for Revised Classification of Epilepsies and Epileptic Syndromes (3).
* History of recent or present significant or medical disease, i.e., cardiovascular, hepatic, renal, gynecologic, musculoskeletal, metabolic, or endocrine.
* History of a severe dermatologic reaction (e.g., Stevens Johnson, toxic epidermolysis necrosis) to medication.
* Subject or parent/legal guardian might not be reasonably expected to be compliant with or to complete the study.
* Participation in a trial of an investigational drug or device within 30 days prior to screening.
* Use of systemic contraceptive for any indication, including acne.

Ages: 30 Months to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 453 (Actual)
Dates: Start 2004-07 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2016-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy A. Glauser, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Peter Adamson, MD, Principal Investigator — Children's Hospital of Philadelphia; Avital Cnaan, PhD, Principal Investigator — Children's National Research Institute
Locations (31):
- United States (31):
  - The Children's Hospital of Alabama, Birmingham, Alabama
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of California at San Diego, La Jolla, California
  - Mattel Children's Hospital at UCLA, Los Angeles, California
  - Children's Hospital of Denver, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nemours Children's Clinic, Jacksonville, Florida
  - Miami Children's Hospital, Miami, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Children's Memorial Hospital, Chicago, Illinois
  - Children's Hospital of Michigan, Detroit, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - Women and Children's Hospital of Buffalo, Buffalo, New York
  - NYU Comprehensive Epilepsy Center, Manhattan, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Rainbow Babies & Children's Hospital, Cleveland, Ohio
  - Children's Hospital, Inc., PCTI, Columbus, Ohio
  - Doernbecher Children's Hospital, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - LeBonheur Children's Medical Center, Memphis, Tennessee
  - Dallas Pediatric Neurology Associates, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Utah/Primary Children's Medical Center, Salt Lake City, Utah
  - Children's Hospital of The King's Daughter (Monarch Medical Research), Norfolk, Virginia
  - Children's Hospital & Regional Medical Center, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Glauser TA, Cnaan A, Shinnar S, Hirtz DG, Dlugos D, Masur D, Clark PO, Adamson PC; Childhood Absence Epilepsy Study Team. Ethosuximide, valproic acid, and lamotrigine in childhood absence epilepsy: initial monotherapy outcomes at 12 months. Epilepsia. 2013 Jan;54(1):141-55. doi: 10.1111/epi.12028. Epub 2012 Nov 21. PMID 23167925
- [Background] Cnaan A, Shinnar S, Arya R, Adamson PC, Clark PO, Dlugos D, Hirtz DG, Masur D, Glauser TA; Childhood Absence Epilepsy Study Group. Second monotherapy in childhood absence epilepsy. Neurology. 2017 Jan 10;88(2):182-190. doi: 10.1212/WNL.0000000000003480. Epub 2016 Dec 16. PMID 27986874
- [Background] Shinnar S, Cnaan A, Hu F, Clark P, Dlugos D, Hirtz DG, Masur D, Mizrahi EM, Moshe SL, Glauser TA; Childhood Absence Epilepsy Study Group. Long-term outcomes of generalized tonic-clonic seizures in a childhood absence epilepsy trial. Neurology. 2015 Sep 29;85(13):1108-14. doi: 10.1212/WNL.0000000000001971. Epub 2015 Aug 26. PMID 26311751
- [Result] Glauser TA, Cnaan A, Shinnar S, Hirtz DG, Dlugos D, Masur D, Clark PO, Capparelli EV, Adamson PC; Childhood Absence Epilepsy Study Group. Ethosuximide, valproic acid, and lamotrigine in childhood absence epilepsy. N Engl J Med. 2010 Mar 4;362(9):790-9. doi: 10.1056/NEJMoa0902014. PMID 20200383
- [Derived] Shinnar RC, Shinnar S, Cnaan A, Clark P, Dlugos D, Hirtz DG, Hu F, Liu C, Masur D, Weiss EF, Glauser TA; Childhood Absence Epilepsy Study Group. Pretreatment behavior and subsequent medication effects in childhood absence epilepsy. Neurology. 2017 Oct 17;89(16):1698-1706. doi: 10.1212/WNL.0000000000004514. Epub 2017 Sep 15. PMID 28916534

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred from July 2004 through October 2007
Groups:
- Ethosuximide: Ethosuximide
  Frequency and Duration: twice a day, every day for the duration of the study treatment
  Formulation: Two formulations were used (actual formulation used was dependent on the patient's weight and ability to swallow): 250mg Zarontin capsules OR 250 mg/5 mL Zarontin syrup
  Dosing: Ethosuximide was titrated in predetermined increments every 1-2 weeks during a 16-week titration period. The titration continued until the patient a) achieved seizure freedom by clinical and EEG criteria, b) reached the maximal allowed study drug dose, c) reached the maximal tolerated dose, or d) developed dose-exiting criteria (treatment failure), whichever came first. Maximum allowed dose: 60 mg/kg/day or 2000 mg/day (whichever was lower)
  Ethosuximide: Ethosuximide is a common treatment for childhood absence epilepsy.
- Lamotrigine: Lamotrigine
  Frequency and Duration: twice a day, every day for the duration of the study treatment
  Formulation: Three formulations were used (actual formulation used was dependent on the patient's weight): 5mg Lamictal chewable tablets OR 25 mg Lamictal chewable tablets OR 25 mg (Lamictal tablets
  Dosing: Lamotrigine was titrated in predetermined increments every 1-2 weeks during a 16-week titration period. The titration continued until the patient a) achieved seizure freedom by clinical and EEG criteria, b) reached the maximal allowed study drug dose, c) reached the maximal tolerated dose, or d) developed dose-exiting criteria (treatment failure), whichever came first. Maximum allowed dose: 12 mg/kg/day or 600 mg/day (whichever was lower).
  Lamotrigine: Lamotrigine is a common treatment for childhood absence epilepsy.
- Valproic Acid: Valproic acid
  Frequency and Duration: twice a day, every day for the duration of the study treatment
  Formulation: Two formulations were used (actual formulation used was dependent on the patient's weight): 250mg Depakote capsules OR 125mg Depakote sprinkles.
  Dosing: Depakote was titrated in predetermined increments every 1-2 weeks during a 16-week titration period. The titration continued until the patient a) achieved seizure freedom by clinical and EEG criteria, b) reached the maximal allowed study drug dose, c) reached the maximal tolerated dose, or d) developed dose-exiting criteria (treatment failure), whichever came first. Maximum allowed dose: 60 mg/kg/day or 3000 mg/day (whichever was lower)
  Valproic acid: Valproic acid is a common treatment for childhood absence epilepsy.
Period: Overall Study
Arm/Group | Ethosuximide | Lamotrigine | Valproic Acid
Started | 156 | 149 | 148
Completed | 155 | 149 | 147
Not Completed | 1 | 0 | 1
Not completed — Did not receive intervention | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ethosuximide | Lamotrigine | Valproic Acid | Total
Number analyzed (Participants) | 155 | 149 | 147 | 451
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 155 | 149 | 147 | 451
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 92 | 76 | 258
  Male | 65 | 57 | 71 | 193
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2
  Asian | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 32 | 26 | 29 | 87
  White | 110 | 117 | 107 | 334
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 12 | 4 | 10 | 26
Region of Enrollment [Number; unit: participants]
  United States | 155 | 149 | 147 | 451
BMI > 90th percentile for age [Count of Participants; unit: Participants] — BMI > 90th percentile for age using the units of kg/m2
  Participants | 43 | 44 | 33 | 120

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Freedom From Treatment Failure at 16-20 Weeks of Double Blind Therapy
Description: Treatment failure was defined as persistence of absence seizures at week 16 or week 20, a generalized tonic-clonic seizure at any time, excessive drug-related systemic toxicity, a moderately severe rash (possibly drug-related), pancreatitis, or increase in the body-mass index of at least 3.0 from baseline, dose-limiting toxicity after a single downward dose modification, or withdrawal initiated by the parent or physician.
Time Frame: First 16-20 weeks of double blind therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Ethosuximide | Lamotrigine | Valproic Acid
Number analyzed (Participants) | 154 | 146 | 146
Participants | 81 | 43 | 85
Statistical Analysis 1: Comparison: Ethosuximide vs Lamotrigine; Calculations of sample size were based on the ability to detect a 20% difference in freedom-from failure rates (three pairwise comparisons) at 16 weeks with 80% power at a two-sided P value of 0.017 and one interim analysis. Sample size of 398 was increased to 446 subjects to account for two stratification factors and a 5% dropout rate; this sample size allowed the detection of a difference of 0.5 SD in the Confidence Index on the Conners' Continuous Performance Test with a power exceeding 80%; Test type: Superiority; p < 0.001, Chi-squared; Odds Ratio (OR) = 2.66, 95% CI 2-sided [1.65 to 4.28] — odds ratio with ethosuximide vs. lamotrigine
Statistical Analysis 2: Comparison: Lamotrigine vs Valproic Acid; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Chi-squared; Odds Ratio (OR) = 3.34, 95% CI 2-sided [2.06 to 5.42] — odds ratio with valproic acid vs. lamotrigine

2. Secondary Outcome: Number of Participants With Attention Deficit as Measured by the Confidence Index of the CPT-II and the K-CPT
Description: A Confidence Index of 0.60 or higher on the Conners' Continuous Performance Test at the visit at 16 or 20 weeks or at an earlier visit when treatment was discontinued (as long as the discontinuation occurred 1 month or more after the baseline visit and was not due to intolerable adverse events). A Confidence Index of 0.60 corresponds to a 60% probability that the child has clinical attention deficit disorder.
Time Frame: First 16-20 weeks of double blind therapy
Population: Those subject who took the Conners' Continuous Performance Test at the visit at 16 or 20 weeks or at an earlier visit when treatment was discontinued (as long as the discontinuation occurred 1 month or more after the baseline visit and was not due to intolerable adverse events).
Measure: Count of Participants; unit: Participants
Arm/Group | Ethosuximide | Lamotrigine | Valproic Acid
Number analyzed (Participants) | 106 | 104 | 106
Participants | 35 | 25 | 52
Statistical Analysis 1: Comparison: Ethosuximide vs Valproic Acid; Test type: Superiority; p = 0.03, Chi-squared; Odds Ratio (OR) = 1.95, 95% CI 2-sided [1.12 to 3.41] — Percentage of subjects with a Confidence Index score of 0.60 or higher in the valproic acid group than in the ethosuximide group
Statistical Analysis 2: Comparison: Lamotrigine vs Valproic Acid; Test type: Superiority; p < 0.001, Chi-squared; Odds Ratio (OR) = 3.04, 95% CI 2-sided [1.69 to 5.49] — Percentage of subjects with a Confidence Index score of 0.60 or higher in the valproic acid group than in the lamotrigine group

3. Secondary Outcome: Number of Participants With Freedom From Treatment Failure at 12 Months of Double Blind Therapy
Description: Treatment failure was defined as persistence of absence seizures at 12 months of double blind therapy, a generalized tonic-clonic seizure at any time, excessive drug-related systemic toxicity, a moderately severe rash (possibly drug-related), pancreatitis, or increase in the body-mass index of at least 3.0 from baseline, dose-limiting toxicity after a single downward dose modification, or withdrawal initiated by the parent or physician.
Time Frame: First 12 months of double blind therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Ethosuximide | Lamotrigine | Valproic Acid
Number analyzed (Participants) | 154 | 146 | 146
Participants | 70 | 31 | 64
Statistical Analysis 1: Comparison: Ethosuximide vs Lamotrigine; Test type: Superiority; p < 0.001, Fisher Exact; Odds Ratio (OR) = 3.08, 95% CI 2-sided [1.81 to 5.33] — Odds ratio for FFF for ethosuximide versus lamotrigine
Statistical Analysis 2: Comparison: Lamotrigine vs Valproic Acid; Test type: Superiority; p < 0.001, Fisher Exact; Odds Ratio (OR) = 2.88, 95% CI 2-sided [1.68 to 5.02] — odds ratio for FFF for valproic acid versus lamotrigine

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over 3.5 years
Description: The definition of adverse event and/or serious adverse event, used to collect adverse event information, is the same as clinicaltrials.gov defintions
Arm/Group | Ethosuximide | Lamotrigine | Valproic Acid
All-Cause Mortality (participants affected / at risk) | 0/155 | 0/149 | 0/147
Serious Adverse Events (participants affected / at risk) | 4/155 | 2/149 | 2/147
Other Adverse Events (participants affected / at risk) | 103/155 | 78/149 | 100/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ethosuximide (N=155) | Lamotrigine (N=149) | Valproic Acid (N=147)
Generalized tonic clonic seizure (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Enteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Due to Salmonella poisoning
Prolonged Absence Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia, diarrhea, vomiting (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Non-epileptic movements (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acting Out (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) — Voluntarily committed
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ethosuximide (N=155) | Lamotrigine (N=149) | Valproic Acid (N=147)
Fatigue (General disorders) | 15 (15) | 13 (13) | 18 (18)
Headache (General disorders) | 19 (19) | 12 (12) | 12 (12)
Sleep problem (General disorders) | 10 (10) | 5 (5) | 14 (14)
Nausea, vomiting, or both (Gastrointestinal disorders) | 23 (23) | 2 (2) | 10 (10)
Stomach upset (Gastrointestinal disorders) | 16 (16) | 4 (4) | 8 (8)
Increased appetite (Gastrointestinal disorders) | 5 (5) | 7 (7) | 13 (13)
Decreased appetite (Gastrointestinal disorders) | 8 (8) | 5 (5) | 3 (3)
Weight increase (Gastrointestinal disorders) | 1 (1) | 3 (3) | 10 (10)
Hyperactivity (Psychiatric disorders) | 14 (14) | 10 (10) | 15 (15)
Hostility (Psychiatric disorders) | 4 (4) | 10 (10) | 18 (18)
Personality change (Psychiatric disorders) | 4 (4) | 9 (9) | 16 (16)
Decrease in concentration (Nervous system disorders) | 6 (6) | 5 (5) | 11 (11)
Somnolence (Nervous system disorders) | 14 (14) | 3 (3) | 4 (4)
Depression (Psychiatric disorders) | 4 (4) | 8 (8) | 8 (8)
Attentional difficulties (Nervous system disorders) | 3 (3) | 5 (5) | 10 (10)
Dizziness (Nervous system disorders) | 9 (9) | 4 (4) | 2 (2)
Memory problems (Nervous system disorders) | 0 (0) | 4 (4) | 8 (8)

LIMITATIONS AND CAVEATS:
This short-term study was not designed to detect long-term systemic or other cognitive effects of these three medications.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Informed Consent Form (2005-08-18): https://cdn.clinicaltrials.gov/large-docs/52/NCT00088452/ICF_000.pdf